CLINICAL TRIAL: NCT01695031
Title: Feasibility of an ED-initiated Online Asthma Management Program for Urban Teens (Puff City-ED)
Brief Title: Feasibility of an ED Initiated Online Asthma Management Program for Urban Teens
Acronym: PuffCityED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: University of Michigan (Other); Children's Hospital of Michigan (Other); Augusta University (Other)
Responsible Party: Principal Investigator, Christine Joseph, Senior Scientist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 1R34HL109296-01A1 (NIH)
Record Dates: First submitted 2012-09-12; First posted 2012-09-27 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Acute Asthma
Keywords: Urban adolescents; Acute asthma; Emergency department; Computer tailoring; Web-based intervention
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tailored asthma management program (Experimental): Teens randomized to the experimental arm will receive 4 sessions of web-based, tailored asthma management
  Interventions: Behavioral: Tailored asthma management program
- Generic web-based education (Active Comparator): Teens in the control group will receive generic, web-based asthma education.
  Interventions: Behavioral: Generic web-based education

INTERVENTIONS:
Behavioral: Tailored asthma management program — web-based, computer-tailored asthma management intervention delivered every week for 4 weeks
  Arms: Tailored asthma management program
Behavioral: Generic web-based education — Generic, web-based asthma education
  Arms: Generic web-based education

SUMMARY:
The objective of this study is to determine the feasibility of conducting a randomized controlled trial to evaluate the effectiveness of an online, Emergency Department-initiated asthma management intervention designed to reduce asthma-related morbidity among urban teenagers aged 13-19 years with uncontrolled asthma. The study will examine issues around recruitment, participant compliance with the study protocol, Internet access, and attrition. Investigators will first develop a protocol for recruiting 13-19 year old patients with acute asthma into an ED-initiated pilot trial of an online asthma management program, describing recruitment and refusal rates. Investigators will measure participant compliance with the pilot study protocol including 4 online sessions and a 6 month survey. Investigators will also measure compliance of the participants parents at baseline and a six month follow up. Investigators will then use pilot study results to describe the intervention effect on selected outcomes including ED visits, asthma control as measured by Asthma Control Questionnaire, functional limitations, quality of life, and behavior change.

DETAILED DESCRIPTION:
Participating emergency departments include Henry Ford Main, Henry Ford Fairlane, and Detroit Medical Center Children's hospital. Eligible teens will be 13-19 years of age. (Including 19 year olds in the the proposed sample means the data is comparable to age categories used by many federal agencies). Eligibility criteria include: a physician diagnosis of acute asthma at the ED visit and parent and teen written informed consent/assent. Eligibility criteria can be confirmed with the help of the ED nursing staff as some teens presenting with symptoms of acute asthma, may receive an asthma diagnosis for the first time in the ED. Using the investigator's data from the school-based trial of Puff City, investigators observed that 12.9% (20/155) of teens reporting an ED visit at baseline also reported no physician diagnosis. This is used as an approximation of the number of participants in the ED pilot that may be newly diagnosed. Teens previously enrolled in the school-based version of Puff City will not be eligible to participate in this pilot. Eligible teens are approached by a recruiter during down time in the ER (while waiting during receiving treatment or while waiting to be discharged). A study recruiter will provide the teen with an enrollment packet that includes an informational brochure (SD 1), a consent (SD 2), and an assent form (SD 3). The recruiter will go through these materials with the parents and teens and answer any questions they may have about the program. The recruited teens who enroll are randomized to either treatment or control. Both groups will be asked to complete an online baseline questionnaire before leaving the ED. An example of this questionnaire has been included with this application (SD 4). Once the baseline questionnaire is finished, teens will then be completing 4 online sessions of web-based asthma education on their own time on a computer with Internet access. Control group will receive commercial websites such as those sponsored by the American Lung Association; the American Academy of Allergy, Asthma and Immunology; the Asthma and Allergy Foundation, and others. Treatment group receives the 4 online, tailored educational sessions. Teens will be encouraged to complete the 4 sessions within 90 days, with a minimum of 7 days between sessions to allow for behavior change. To regulate dosage, control participants receive a "time expired" message after 30 minutes of browsing; this time limit is commensurate with the estimated time needed to complete a tailored session. Teens will also be asked to complete a 6-month follow-up survey (SD 5).Parents/Guardians of the enrolled teens will also be asked to complete a baseline questionnaire and a follow-up at 6 months (SD 6-7) in the form of a telephone interview with a trained interviewer.

In YR1 investigators will develop the recruitment protocol, hire and train recruiters, and establish a study database. Investigators will get on the agenda of CHM ED staff meetings to orient clinic staff to the intervention, obtain input/feedback, discuss logistics, address concerns, and answer questions about the project. Prior to recruitment Investigators will develop signage about the study (as appropriate) for the ED. Recruitment will start in month six of YR1, with at least two practice runs of the protocol. In YR2, investigators will continue recruitment and begin 6 month follow-up surveys. Recruitment will end in the fall of YR2 leaving 6-8 months for completion of follow-up, analysis and write-up. At the end of YR1 and again at the end of YR2, investigators will conduct short, qualitative interviews with ED and research staff to ensure identification of issues, barriers, and obstacles to conducting a trial of an ED-initiated version of Puff City.

ELIGIBILITY:
Inclusion Criteria:

* 13-19 years of age
* Physician diagnosis of acute asthma at the Emergency Department visit
* Parent written informed consent
* Teen written informed assent

Exclusion Criteria:

* Inability to provide informed consent/assent
* No physician diagnosis of asthma
* Other co-morbidities that make it impossible for individual to participate.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Emergency Department Visit | 12 months
  Proportion of enrolled teens randomized to the treatment group who return to the ED with acute asthma compared to the proportion of enrolled teens randomized to the control group who return to the ED with acute asthma

SECONDARY OUTCOMES:
Asthma Control Test (ACT) | 12 months
  Comparison of ACT scores at 12 months post-baseline by randomization group

OTHER OUTCOMES:
Functional Status | 12 months
  Compare functional status (e.g., symptom-days, symptom-nights, days of restricted activity, school/work days missed, etc.) by randomization group at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine LM Joseph, PhD, MPH, Principal Investigator — Henry Ford Health System
Locations (2):
- United States (2):
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan

REFERENCES:
- [Derived] Joseph CLM, Mahajan P, Stokes-Buzzelli S, Johnson DA, Duffy E, Williams R, Zhang T, Ownby DR, Considine S, Lu M. Pilot study of a randomized trial to evaluate a Web-based intervention targeting adolescents presenting to the emergency department with acute asthma. Pilot Feasibility Stud. 2017 Jun 21;4:5. doi: 10.1186/s40814-017-0147-6. eCollection 2018. PMID 28649417